CLINICAL TRIAL: NCT07303517
Title: ACCESS: AI-Driven Consent Simplification Study
Brief Title: AI-Driven Consent Simplification Study
Acronym: ACCESS
Status: Not yet recruiting | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Other Study IDs: IRB-24-6074
Record Dates: First submitted 2025-12-08; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Informed Consent; Comprehension; Communication; Disclosure
Keywords: Informed Consent Readability; Plain language; Simplified consent forms; Research ethics
MeSH Terms: conditions — Communication

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Group 1-Adult participants - Arm A: Will review the original ICF
  Interventions: Behavioral: Original ICF
- Group 1 - Adult participants - Arm B: Will review the simplified ICF
  Interventions: Behavioral: AI Simplified ICF
- Group 1- Adult participants - Arm C: Will listen to a podcast in conjunction to the original ICF
  Interventions: Behavioral: Original ICF; Behavioral: Podcast - Original ICF
- Group 1-Adult participants - Arm D: Will listen to a podcast in conjunction to the simplified ICF
  Interventions: Behavioral: AI Simplified ICF; Behavioral: Podcast - Simplified ICF
- Group 2 - Investigators: PIs who are health providers that perform clinical trials
  Interventions: Behavioral: Original ICF; Behavioral: AI Simplified ICF; Behavioral: Podcast - Original ICF
- Group 3 - IRB individuals: Individuals involved in IRB activities (chairs, committee members, staff)
  Interventions: Behavioral: Original ICF; Behavioral: AI Simplified ICF; Behavioral: Podcast - Original ICF

INTERVENTIONS:
Behavioral: Original ICF — Participant will review the original ICF
  Groups: Group 1- Adult participants - Arm C; Group 1-Adult participants - Arm A; Group 2 - Investigators; Group 3 - IRB individuals
Behavioral: AI Simplified ICF — Participant will review the AI Simplified ICF
  Groups: Group 1 - Adult participants - Arm B; Group 1-Adult participants - Arm D; Group 2 - Investigators; Group 3 - IRB individuals
Behavioral: Podcast - Original ICF — Listen to a podcast that is developed to provide an engaging format for the original ICF.
  Groups: Group 1- Adult participants - Arm C; Group 2 - Investigators; Group 3 - IRB individuals
Behavioral: Podcast - Simplified ICF — Listen to a podcast that is developed to provide an engaging format for the simplified ICF.
  Groups: Group 1-Adult participants - Arm D

SUMMARY:
The overarching goal of this pilot is to explore how generative artificial intelligence (genAI) can be used to improve the accessibility and understandability of informed consent materials in clinical research. The study will test the extent to which informed consent text can be improved by large language models (LLM; specifically, ChatGPT and NotebookLM) along with other AI tools (specifically, ElevenLabs) through qualitative and quantitative analyses.

Simplifying such forms using genAI may facilitate better comprehension, ensuring truly informed consent. Improving informed consent form (ICF) comprehension can lead to more informed and willing participation in clinical studies. This improved understanding may result in higher enrollment rates, better subject retention, and more accurate data collection as individuals will have a clearer understanding of study procedures and risks.

ELIGIBILITY:
Inclusion Criteria:

Group 1:

* Age 60 years and above
* UCLA patient
* English speaking
* Ability to provide informed consent

Group 2:

* UCLA investigators who are health providers that perform clinical trials
* Must be clinical research investigatory and staff actively involved in research operations at UCLA
* English speaking

Group 3:

* Individuals involved in IRB activities (chairs, committee members, staff)
* Must be a director or staff at UCLA
* English speaking

Exclusion Criteria:

* Group 1: None
* Group 2: PI and co-PIs of the study "Donor Chimerism and Graft Survival Following Combined HLA-Identical Sibling Living Donor Kidney and Hematopoietic Stem Cell Transplantation Utilizing a Conditioning Regimen of Total Lymphoid Irradiation (TLI) and Rabbit Anti-Thymocyte Globulin (rATG)"
* Group 3: Individuals from the IRB who have reviewed the study submission for "Donor Chimerism and Graft Survival Following Combined HLA-Identical Sibling Living Donor Kidney and Hematopoietic Stem Cell Transplantation Utilizing a Conditioning Regimen of Total Lymphoid Irradiation (TLI) and Rabbit Anti-Thymocyte Globulin (rATG)"

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: UCLA patients, principal investigators (PIs) and institutional review board (IRB) members will be enlisted to evaluate 1 of the ICFs. Patient cohort will be identified using the Mental Health and Smart Technology Registry, The Diabetes Research Registry, and/or the EMBRACE registry and contacted by email. The PI cohort will be identified by direct referrals.
Sampling Method: Non-Probability Sample
Enrollment: 230 (Estimated)
Dates: Start 2026-01-08 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Quality of Informed Consent (QUIC) | Day 1 (immediately after reviewing the ICF materials)
  The QUIC measures knowledge recall. The summed score of 10 knowledge items comprising key concepts of informed consent will be calculated. The scores range between 0 and 22 with higher scores indicating higher knowledge.

SECONDARY OUTCOMES:
Time to read and understand informed consent | Day 1
  The time taken by each participant to complete reading and understanding of the ICF materials.
Participant understanding and comprehension of the study | Day 1
  10-15 questions specific to the ICF and the study protocol

CONTACTS AND LOCATIONS:
Overall Officials: Arash Naeim, MD, PhD, Principal Investigator — University of California, Los Angeles

IPD SHARING:
Plan to Share IPD: No